CLINICAL TRIAL: NCT01300273
Title: Phase 4 Study of Mechanisms of Low Protein Diet Supplemented With Ketoanalogs on Reducing Proteinuria and Maintaining Nutritional Status in Type 2 Diabetic Nephropathy
Brief Title: Low Protein Diet Supplemented With Ketoanalogs on Reducing Proteinuria and Maintaining Nutritional Status in Type 2 Diabetic Nephropathy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Collaborators: Huashan Hospital (Other); Shanghai East Hospital (Other); Shanghai 6th People's Hospital (Other)
Responsible Party: Principal Investigator, Weijie Yuan, Chief physician, Director of Department of Nephrology, Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KETO-011-IP4
Record Dates: First submitted 2011-02-18; First posted 2011-02-21 (Estimated); Last update posted 2011-09-08 (Estimated); Status verified 2011-09

CONDITIONS: Type 2 Diabetic Nephropathy
Keywords: Diabetic nephropathy; Podocyte; Low Protein Diet; Ketoanalogs
MeSH Terms: conditions — Diabetic Nephropathies | interventions — ketosteril

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ketosteril (Experimental)
  Interventions: Dietary Supplement: Compound α-Ketoacid Tablet

INTERVENTIONS:
Dietary Supplement: Compound α-Ketoacid Tablet — 30 patients will be treated with a LPD containing 0.6g protein/kg BW per day and 120-125 kJ/kg BW per day and supplemented with keto-amino acids (Ketosteril®, Fresenius Kabi) at a dosage of 100 mg/kg BW per day.
  Other Names: Ketosteril; Ketoanalogs

SUMMARY:
The investigators hypothesize that, LPD supplemented with ketoanalogs will reduce urine podocyte loss and lower the angiotensinogen level in the urine.

DETAILED DESCRIPTION:
Diabetic nephropathy is one of the most important causes of end stage renal disease in the world. Recently In a multicenter, randomized clinical trial performed in China, which aimed to evaluate the efficacy and safety of compound α-keto acid tablet in combination with low protein diet (LPD+KA) in delaying the progress of type 2 diabetic nephropathy(T2DN). In that study it was found that LPD+KA was associated with amelioration of proteinuria, better reduction in the loss of kidney function compared with LPD alone meanwhile nutrition status remained well in both group(Role of Ketoanalogs in diabetic nephropathy-China study, to be submitted for publication). However, in that study the mechanisms underlined these effects were not been elucidated This research proposal is a part of the continuation of that study. Restriction of Protein intake, strictly control blood pressure, particularly using renin-angiotensin system (RAS) blockade have been shown to ameliorate proteinuria and progression of CKD. Podocyte damage has been know to play critical role for proteinuria and renal function loss A recent study showed that the mRNA expression of podocyte markers in urinary sediment is increased in patients with T2DN, and this effect can be inhibited by ACE inhibitor and ARB, which indicates the important role of local renal RAS to involve in the damage. Urinary angiotensinogen level is a good marker of the situation of renal RAS. Consequently the investigators are proposing to study the effect of LPD+KA on podocyte as well as on local RAS in the kidney.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with type 2 diabetes
* age range is 18 - 80 years old
* no gender restrictions
* use oral hypoglycemic agents (limited to repaglinide, α-glucosidase inhibitor and chloroquine ketone) and/or insulin to control blood sugar
* fasting blood sugar is not higher than 10mmol/l, glycated hemoglobin is not higher than 8.5%
* using RAS system blockers (ACEI or ARB) for at least 4 weeks and blood pressure is no higher than 160/90mmHg. Once enrolled in the group, the dose should not be changed, unless there is contraindication
* has not yet started dialysis, GFR based on simplified MDRD formula is between (15-60) ml/min/1.73m2
* serum albumin is not less than 25g/l and appearing dominant proteinuria (urinary albumin excretion rate > 300mg/24h)
* understanding and willing to participate in the trial and signed informed consent

Exclusion Criteria:

* compliance is poor
* GFR < 15ml/min/1.73m2
* repeated hypercalcemia, hyperkalemia
* ketoacidosis occurred in recent 6 months
* chronic heart failure, above NYHA 3 grade
* combined with other serious diseases in 3 months
* obvious symptoms and signs of liver disease. Alanine or aspartate aminotransferase 2 times higher than normal
* severe edema, or up to the level of nephrotic syndrome or that there is serous cavity effusion
* urinary tract infections or other urinary tract diseases
* drug abusers
* diagnosed of malignancy
* receiving long-term systemic steroid therapy
* women pregnancy or Intended pregnancy and breastfeeding
* took part in other clinical drug studies 30 days before the trial

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2011-02; Primary Completion 2012-05 (Estimated); Study Completion 2012-07 (Estimated)

PRIMARY OUTCOMES:
monitor podocyte loss by detecting nephrin, podocin, and synaptopodin mRNA in urine particulates with quantitative reverse transcriptase-PCR. | At baseline and every 3 months
  At baseline and every 3 months, a whole-stream early morning urine specimen will be collected for gene expression study.

CONTACTS AND LOCATIONS:
Overall Officials: Weijie Yuan, Professor, Principal Investigator — Department of Nephrology, First People's Hospital, Shanghai Jiao Tong University
Locations (1):
- Department of Nephrology,Shanghai Jiaotong University Affiliated First People's Hospital, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Background] Kasiske BL, Lakatua JD, Ma JZ, Louis TA. A meta-analysis of the effects of dietary protein restriction on the rate of decline in renal function. Am J Kidney Dis. 1998 Jun;31(6):954-61. doi: 10.1053/ajkd.1998.v31.pm9631839.
- [Background] Mahmood J, Khan F, Okada S, Kumagai N, Morioka T, Oite T. Local delivery of angiotensin receptor blocker into the kidney ameliorates progression of experimental glomerulonephritis. Kidney Int. 2006 Nov;70(9):1591-8. doi: 10.1038/sj.ki.5001872. Epub 2006 Sep 20. PMID 16985512
- [Background] Wang G, Lai FM, Lai KB, Chow KM, Li KT, Szeto CC. Messenger RNA expression of podocyte-associated molecules in the urinary sediment of patients with diabetic nephropathy. Nephron Clin Pract. 2007;106(4):c169-79. doi: 10.1159/000104428. Epub 2007 Jun 26. PMID 17596726
- [Background] Wang G, Lai FM, Lai KB, Chow KM, Kwan BC, Li PK, Szeto CC. Urinary messenger RNA expression of podocyte-associated molecules in patients with diabetic nephropathy treated by angiotensin-converting enzyme inhibitor and angiotensin receptor blocker. Eur J Endocrinol. 2008 Mar;158(3):317-22. doi: 10.1530/EJE-07-0708. PMID 18299464
- [Background] Yamamoto T, Nakagawa T, Suzuki H, Ohashi N, Fukasawa H, Fujigaki Y, Kato A, Nakamura Y, Suzuki F, Hishida A. Urinary angiotensinogen as a marker of intrarenal angiotensin II activity associated with deterioration of renal function in patients with chronic kidney disease. J Am Soc Nephrol. 2007 May;18(5):1558-65. doi: 10.1681/ASN.2006060554. Epub 2007 Apr 4. PMID 17409316
- [Background] Adey D, Kumar R, McCarthy JT, Nair KS. Reduced synthesis of muscle proteins in chronic renal failure. Am J Physiol Endocrinol Metab. 2000 Feb;278(2):E219-25. doi: 10.1152/ajpendo.2000.278.2.E219. PMID 10662705
- [Background] Sato N, Komatsu K, Kurumatani H. Late onset of diabetic nephropathy in spontaneously diabetic GK rats. Am J Nephrol. 2003 Sep-Oct;23(5):334-42. doi: 10.1159/000072915. Epub 2003 Aug 13. PMID 12920324
- [Background] Verity MA. Infantile Pompe's disease, lipid storage, and partial carnitine deficiency. Muscle Nerve. 1991 May;14(5):435-40. doi: 10.1002/mus.880140509. PMID 1870635